CLINICAL TRIAL: NCT06709560
Title: Sex Differences in Baroreflex Sensitivity Response to Different Constant-load Submaximal Exercise Intensities
Brief Title: Baroreflex Sensitivity Response to Exercise
Acronym: PACE MAKERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Faculdade de Motricidade Humana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PACE MAKERS
Record Dates: First submitted 2024-11-23; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Sex
Keywords: Hear Rate Variability; Baroreflex Sensitivity; Exercise Intensity; Acute Exercise; Sex Differences
MeSH Terms: conditions — Coitus | interventions — Blood Pressure

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were blinded to the order of the visits until arrival at the laboratory.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heart Rate Reserve (HRR)-Based Exercise Intensity Prescription (Active Comparator): The exercise intensity is based solely on HRR.
  Interventions: Other: Moderate Intensity Continuous Exercise; Other: Vigorous Intensity Continuous Exercise
- Blood Pressure-Matched Exercise Intensity Prescription (Experimental): Instead of relying on HRR, exercise intensity is tailored to replicate the average systolic blood pressure achieved in the initial HRR-based session.
  Interventions: Other: Moderate Intensity Continuous Exercise Matched for Blood Pressure; Other: Vigorous Intensity Continuous Exercise Matched for Blood Pressure

INTERVENTIONS:
Other: Moderate Intensity Continuous Exercise — Participants perform a continuous cycling exercise session on a reclined ergometer at moderate intensity (50% HRR)
  Arms: Heart Rate Reserve (HRR)-Based Exercise Intensity Prescription
Other: Vigorous Intensity Continuous Exercise — Participants perform a continuous cycling exercise session on a reclined ergometer, at a vigorous intensity (80% HRR).
  Arms: Heart Rate Reserve (HRR)-Based Exercise Intensity Prescription
Other: Moderate Intensity Continuous Exercise Matched for Blood Pressure — Participants perform a cycling session where exercise intensity is adjusted to match the systolic blood pressure levels attained during the first visit at moderate intensity (50% HRR).
  Arms: Blood Pressure-Matched Exercise Intensity Prescription
Other: Vigorous Intensity Continuous Exercise Matched for Blood Pressure — Participants perform a different cycling session where exercise intensity is adjusted to match the systolic blood pressure levels attained during the first visit at vigorous intensity (80% HRR).
  Arms: Blood Pressure-Matched Exercise Intensity Prescription

SUMMARY:
Males and females show distinct differences in cardiovascular function, especially during exercise. Evidence suggests that females generally have lower blood pressure due to hormonal influences that reduce blood vessel constriction. This protective effect may contribute to a lower risk of high blood pressure and cardiovascular diseases in females compared to males. Additionally, females tend to have different patterns of heart rate control and blood pressure regulation, largely due to differences in the autonomic nervous system and hormonal balance.

One key mechanism involved in blood pressure control is the baroreflex, which helps stabilize blood pressure by adjusting heart rate and blood vessel function. The sensitivity of the baroreflex (known as baroreflex sensitivity, or BRS) can vary between males and females. For instance, females may exhibit slower adjustments in heart rate in response to blood pressure changes, but they also tend to have better blood pressure regulation during moderate exercise.

The main purpose of this study is to explore whether these sex-specific differences extend to more intense exercise. Investigators will compare the responses of young, active males and females to cycling at two exercise intensities: moderate (50% of Heart Rate Reserve, HRR) and vigorous (80% HRR). As a secondary purpose, investigators we will assess the inter-day repeatability of HRV and BRS parameters measured at rest and during moderate and vigorous intensity exercise utilizing sequence and spectral indices in apparently healthy young adult males and females.

We hypothesize that:

1. Females will show higher HRV and BRS at rest compared to males, indicating better heart rate control.
2. During exercise, females will have greater cardiovagal (heart-related) activation than males, regardless of exercise intensity.
3. When exercise sessions are matched for blood pressure, there will be no significant sex differences in HRV and BRS responses.
4. Sequential methods techniques can be used to assess cardiovagal BRS and HRV changes between days during exercise in young adults, regardless of their sex. In addition, the inclusion of vigorous intensity may improve the repeatability of the outcome measure due to sympathetic outflow predominance.

DETAILED DESCRIPTION:
Forty healthy and physically active participants (20 males and 20 females) aged 18-31 were recruited for this study. All participants reported to the laboratory in a fasted state (>4 hours) and refrained from consuming foods or drinks containing caffeine or alcohol for at least 12 hours. They also avoided strenuous exercise for at least 24 hours prior to the testing sessions. The menstrual cycle was not controlled for female participants. All participants provided written informed consent after receiving a detailed explanation of the study's aims and experimental procedures.

This study was constructed as a crossover trial. Participants attended 4 separate intervention sessions. On the first visit, participants had their body composition evaluated by a clinical bioimpedance device using 8 electrodes positioned on each hand and foot. Each participant also performed a ramp incremental cycle ergometer test to exhaustion on a recumbent stationary cycle ergometer (Excite Recline Med, TechnoGym, Italy). On the second and third visit, participants quietly rested for 15 min in the supine position to evaluate heart rate variability (HRV) using a 5-ECG lead module (Nova, Finapres Measurement Systems, Amsterdam, The Netherlands), carotid (Arietta V60 ultrasound; Aloka/Hitachi Medical Systems) and aortic (Complior Analyse software (ALAM Medical, Paris, France) arterial stiffness. Participants then performed a 6 minutes bout of moderate intensity continuous exercise (MICE) at 50% heart rate reserve [HRR= 0.5*(HRmax- HRrest) + HRrest] followed by a 6 minutes vigorous intensity continuous exercise (VICE) bout at 80% HRR on a recumbent stationary bike, while having their HRV, beat-by-beat blood pressure and carotid arterial stiffness evaluated at HR steady state at each intensity. Visits 2 and 3 provided the data for the repeatability objective and hypothesis. On the fourth visit, the participants performed an acute bout of MICE and VICE, but this time at the corresponding average blood pressure at each intensity from visits 2 and 3. As men show higher blood pressure values during exercise, in the fourth visit we matched their intensity of exercise with the average blood pressure attained by women during steady state at each intensity.

Blood pressure and HR were monitored beat-by-beat and carotid arterial stiffness was measured at BP steady-state.

All visits were conducted in the morning with each participant performing sessions at the same time of the day to minimize any potential diurnal variation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 44 years old.
* Physical active as assessed by the International Physical Activity Questionnaire (IPAQ).
* Low risk to increase physical Activity as assessed by the Physical Activity Readiness Questionnaire (PAR-Q+).

Exclusion Criteria:

* Smoking
* Diagnosed with cardiac, metabolic or renal diseases
* Taking cardioactive medication
* Resting hypertension (systolic blood pressure >140 mmHg, diastolic blood pressure > 90 mmHg).

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Changes in Heart Rate Variability | At rest and in the last 2 minutes of the 6 minutes bout of MICE and VICE
  R-R intervals were derived from beat-to-beat blood pressure pulse intervals using finger plethysmography (Finapres® Nova, Amsterdam, Netherlands) at rest and during exercise across all visits. The pressure signal's upstroke was identified with a 2 ms resolution, and the interval between consecutive upstrokes was measured. In the frequency domain, low-frequency (LF; 0.04-0.15 Hz) reflected sympathetic and parasympathetic modulation, while high-frequency (HF; 0.15-0.40 Hz) served as a marker of parasympathetic modulation. The LF/HF ratio indicated sympathovagal dominance. Data acquisition and analysis were conducted following the Task Force guidelines of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology.
Changes in Baroreflex sensitivity | At rest and in the last 2 minutes of the 6 minutes bout of moderate intensity continuous exercise and high intensity continuous exercise
  A spectral method was used to compute baroreflex sensitivity as the transfer gain of the cross-spectra between pressure and interval at rest and during exercise across all visits. Coherence was typically high in the 10 s rhythm band (0.06-0.15 Hz) and at ventilatory frequencies (0.15-0.5 Hz). Spectral estimates of the recordings were computed using the Finapres® Nova device software (Amsterdam, Netherlands), which provided an easy-to-use interface. A discrete Fourier transform, requiring no interpolation or zero padding, was applied. Triangular spectral smoothing was set at a width of 10, reflecting the 10-minute duration of the recordings. Spectral density, coherence, pressure-interval transfer gain, and phase plots were displayed on the device screen, with a cursor allowing manual selection of bands with high coherence and spectral power. An output program listed the resultant data and all selections made for subsequent analysis.

SECONDARY OUTCOMES:
Regional Arterial Stiffness | At rest in each visit to the laboratory, just before the 6 minutes bouts of MICE and VICE
  Arterial stiffness was measured by pulse wave velocity (PWV) using applanation tonometry. The distance between the carotid and femoral arteries was measured directly and entered into the Complior Analyse software (ALAM Medical, Paris, France) with a correction factor of 0.8. Right brachial blood pressure was measured twice and entered into the software before initiating signal acquisition. The operator positioned the carotid sensor using its holder and manually held the femoral and distal posterior tibial sensors. When 10 high-quality carotid pulse waveforms were observed, simultaneous carotid and femoral pressure curves were recorded for 10 pulse waveforms. The transit time between the two waveforms was automatically calculated. Values from the carotid to femoral artery were used as an index of central/aortic arterial stiffness.
Central Blood Pressure | At rest and in the last 2 minutes of the 6 minutes bout of moderate intensity continuous exercise and high intensity continuous exercise
  Carotid Systolic Blood Pressure (SBP) was assessed from right carotid traces acquired by applanation tonometry (Complior Analyse). The waveforms were averaged, and the mean values will be extracted from 15 s window of acquisition. The carotid waveforms were calibrated from MAP and brachial SBP, measured immediately before the acquisition.
Changes in Local Arterial Stiffness | At rest and in the last 2 minutes of the 6 minutes bout of moderate intensity continuous exercise and high intensity continuous exercise
  Carotid arterial stiffness indices were assessed using eTRACKING technology. Common carotid diameter values and diameter-derived pressure data calculated Peterson's pressure-strain elastic modulus (ε) and stiffness index (β) using published algorithms. The augmentation index (AIx), reflecting arterial wave reflection, was calculated as the ratio of augmented pressure (difference between the carotid pressure curve "shoulder" and peak systolic pressure) to pulse pressure. AIx was derived using the third derivative method to locate the pulse inflection point. Measurements were performed at rest and during exercise across all visits.
Changes in Carotid Blood Pressure Wave Intensity | At rest and in the last 2 minutes of the 6 minutes bout of moderate intensity continuous exercise and high intensity continuous exercise
  Wave intensity was calculated as the product of the derivatives of simultaneously recorded blood pressure and blood flow velocity changes, obtained at specific circulatory points. Blood pressure waveforms were derived non-invasively using a system developed by Hitachi, leveraging the correlation between cyclic blood pressure and vessel diameter changes.
  The right common carotid artery was scanned using an Arietta V60 ultrasound machine (Hitachi Aloka Medical Ltd, Mitaka-shi, Tokyo, Japan) with a 7.5 MHz linear probe and a 5 MHz Doppler transducer at rest and during exercise. The intima-media borders were tracked using high-resolution wall tracking at 1 kHz. Arterial pressure waveforms were calibrated with sphygmomanometry, and flow velocity was recorded using Doppler ultrasound. Data were averaged from approximately 20 beats to derive waveforms and net wave intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Ginásio Clube Português, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Data obtained in this study may be provided to qualified researchers with academic interest in the effects of acute exercise on the autonomic function. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact xmelo@egasmoniz.edu.pt

REFERENCES:
- [Background] Bassareo PP, Crisafulli A. Gender Differences in Hemodynamic Regulation and Cardiovascular Adaptations to Dynamic Exercise. Curr Cardiol Rev. 2020;16(1):65-72. doi: 10.2174/1573403X15666190321141856. PMID 30907327
- [Background] Seo MW, Park TY, Jung H. Sex Differences in Heart Rate Variability and Vascular Function Following High-Intensity Interval Training in Young Adults. J Hum Kinet. 2023 Oct 11;90:89-100. doi: 10.5114/jhk/170964. eCollection 2024 Jan. PMID 38380301
- [Background] Schumann A, Gupta Y, Gerstorf D, Demuth I, Bar KJ. Sex differences in the age-related decrease of spontaneous baroreflex function in healthy individuals. Am J Physiol Heart Circ Physiol. 2024 Jan 1;326(1):H158-H165. doi: 10.1152/ajpheart.00648.2023. Epub 2023 Nov 10. PMID 37947436
- [Background] Wheatley CM, Snyder EM, Johnson BD, Olson TP. Sex differences in cardiovascular function during submaximal exercise in humans. Springerplus. 2014 Aug 20;3:445. doi: 10.1186/2193-1801-3-445. eCollection 2014. PMID 25191635
- [Background] Fu Q, Ogoh S. Sex differences in baroreflex function in health and disease. J Physiol Sci. 2019 Nov;69(6):851-859. doi: 10.1007/s12576-019-00727-z. Epub 2019 Nov 12. PMID 31721084